CLINICAL TRIAL: NCT06322212
Title: Type 2 Diabetes Mellitus and Blood Brain Barrier Improvement - A Randomized Clinical Trial
Brief Title: Type 2 Diabetes and Blood Brain Barrier Improvement
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rajesh Kumar, PhD, Professor of Anesthesiology and Radiological Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-001083; 1R21AG085268-01 (NIH)
Record Dates: First submitted 2024-03-07; First posted 2024-03-20 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Type2diabetes
Keywords: MRI; Thiamine Treatment; Thiamine Deficiency; Cognition Assessments
MeSH Terms: conditions — Thiamine Deficiency | interventions — Thiamine

STUDY DESIGN:
Intervention Model Description: Compare BBB function, cognition, and mood in T2DM adults with and without Thiamine treatment.
Who Masked: Participant
Masking Description: Participants will be assigned a number to be used instead of their names with double-blind randomization until visits are complete and data is analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BBB function, cognition, and mood in T2DM adults with Thiamine treatment. (Experimental): Analyze BBB function, cognition, and mood in T2DM adults with Thiamine treatment and compare to the placebo group.
  Interventions: Dietary Supplement: Thiamine
- BBB function, cognition, and mood in T2DM adults without Thiamine treatment. (Placebo Comparator): Analyze BBB function, cognition, and mood in T2DM adults without Thiamine treatment and compare to the Thiamine treatment group.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Thiamine — Participants will be provided instruction to take one 500 mg capsule of Thiamine (Vitamin B1) each day in the morning for 3-months.
  Other Names: B1
  Arms: BBB function, cognition, and mood in T2DM adults with Thiamine treatment.
Other: Placebo — Participants will be provided instruction to take one capsule (placebo) each day in the morning for 3-months.
  Other Names: inactive
  Arms: BBB function, cognition, and mood in T2DM adults without Thiamine treatment.

SUMMARY:
The majority of T2DM adults show thiamine (vitamin B1) deficiency which may contribute to impaired function. This study will examine patients with T2DM through brain MRI scans, cognition assessments, blood tests, and questionnaires. Our goal is to see if a thiamine treatment (taking vitamin B1 capsules) can improve function. Patients will be asked to come to UCLA two times three months apart and each visit will last about 2.5-3 hours.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) makes up 90-95% of all diagnosed diabetes mellitus, and is a serious health issue in the United States.1 T2DM adults show significant mood and cognitive deficits, symptoms that are associated with higher morbidity and mortality, poor self-care, and decreased quality of life, and the condition is linked with early dementia and Alzheimer's disease. Brain structural changes emerge in T2DM adults in sites that exert major influence on cognition and mood functions, potentially resulting from impaired blood brain barrier function (BBB). However, it is unclear whether BBB function can be repaired in T2DM adults, reducing impaired cognition and mood functions and early risks of dementia and Alzheimer's disease in the condition.

Several pre-clinical studies suggest the possibility for BBB function repair, including low-cost thiamine intervention. Thiamine is an essential co-factor for carbohydrate metabolism and adequate or higher levels promote aerobic metabolism and reduce neural injury. In addition, reduced thiamine levels are shown contributing to impaired endothelial cell functions and higher doses of thiamine treatment improve endothelial functions. Thus, lower thiamine levels can contribute to neural, as well as endothelial cell dysfunctions, resulting to impaired BBB function. The majority of T2DM adults show thiamine deficiency, which may contribute to impaired BBB function, but it is unclear if the thiamine treatment can improve BBB function in T2DM adults. The investigators hypothesize that thiamine intervention (3-months) will reduce impaired BBB function and will improve cognition and mood functions in T2DM adults with thiamine treatment compared to non-treated T2DM adults.

In summary, the investigators propose that low-cost thiamine treatment for 3-months in T2DM adults will repair BBB dysfunction and improve mood and cognition functions. If studies successful, the findings from this clinical trial might serve as a novel and innovative treatment strategy to repair BBB function, affecting less cognition and mood function, and hence better outcomes in T2DM adults, as well as in other adult conditions with impaired BBB function. This R21 exploratory clinical trial study will provide required data regarding the benefits of a low-cost thiamine intervention that could be implemented on a large-scale clinical trial to repair BBB function in T2DM adults, as congruent to the National Institutes of Health mission, and thus, decrease early risks of dementia and Alzheimer's disease, reduce morbidity and mortality, and increase quality of life in this serious and common T2DM patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed T2DM
* Outpatient status
* Able to lay flat for imaging

Exclusion Criteria:

* A previous history of stroke
* Current in-take of thiamine
* Known thiamine allergy
* Seizure disorder
* Head trauma
* Myocardial infarction
* Current pregnancy (if female)
* Diagnosed neuropsychiatric disorders (clinical depression, schizophrenia, manic-depression)
* Diagnosed dementia
* Sleep disordered breathing
* Airway or chest deformities that would interfere with breathing
* Chronic obstructive pulmonary disease
* Cystic fibrosis
* Presence of brain mass lesions
* Any history of drug abuse (e.g., cocaine, tobacco, or cannabis)
* Renal failure (requiring dialysis)
* All T2DM adults with metallic and electronic implants (phrenic or cardiac pacemakers; although some pacemakers and cardioverter defibrillators are safe at a low magnetic field, they are not safe at 3.0-Tesla scanner)
* Non-removable insulin pump/glucose sensor
* Braces
* Body weight more than 300 pounds (weight and height will be used to calculate BMI to determine if the patient will fit in the scanner and stay within parameters of size restrictions of MRI scanner table)
* Any other contraindications to MRI, such as claustrophobia, or metallic-based tattoos, as per MRI safety website suggestions, will also be excluded.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Assess if BBB function has been repaired. | After 3 months
  Assess the function of the Blood Brain Barrier.
Analyze blood serum S100β levels. | After 3 months
  Analyze blood serum S100β (marker of BBB integrity) levels to see if they have been reduced in thiamine treated T2DM adults over T2DM adults without thiamine treatment.
Examine cognition in T2DM adults with thiamine treatment. | After 3 months
  The investigator will examine cognition using the Wide Range Assessment of Memory and Learning 2 (WRAML2) to see if T2DM adults with thiamine treatment show improved cognition over T2DM adults without thiamine treatment.
Cognition assessment in T2DM adults after thiamine treatment. | After 3 months
  The investigator will assess cognition using the Montreal Cognitive Assessment (MoCA) to see if T2DM adults with thiamine treatment show improved cognition over T2DM adults without thiamine treatment.
Examine depression in T2DM adults with thiamine treatment. | After 3 months
  The investigator will examine depression using using the Beck Depression Inventory II (BDI-II) to see if T2DM adults with thiamine treatment have an improvement in mood compared to T2DM adults without thiamine treatment.
Assess anxiety in T2DM adults with thiamine treatment. | After 3 months
  The investigator will assess anxiety using using the Beck Anxiety Inventory (BAI) to see if T2DM adults with thiamine treatment have an improvement in mood compared to T2DM adults without thiamine treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigator will make every effort to publish data in a timely manner. Once the findings related to changes in blood brain barrier based on brain MRI data before and after thiamine intervention have been published or by the end of award performance period, whichever is sooner, the MRI data, demographics, mood and cognition, and clinical data (devoid of individual identifiers) will be deposited in NIH supported domain-specific data sharing repository (NIMH Data Archive). All data will be labeled with consistent unique identifiers that will make it easily findable in data repository to interested research investigators. Data will be available forever after sharing with data repository to other investigators for secondary analyses.
Supporting Information: CSR
Time Frame: Once the findings related to changes in blood brain barrier based on brain MRI data before and after thiamine intervention have been published or by the end of award performance period, whichever is sooner.
Access Criteria: Any research investigator

REFERENCES:
- [Background] Umegaki H. Type 2 diabetes as a risk factor for cognitive impairment: current insights. Clin Interv Aging. 2014 Jun 28;9:1011-9. doi: 10.2147/CIA.S48926. eCollection 2014. PMID 25061284
- [Background] Vincent C, Hall PA. Executive Function in Adults With Type 2 Diabetes: A Meta-Analytic Review. Psychosom Med. 2015 Jul-Aug;77(6):631-42. doi: 10.1097/PSY.0000000000000103. PMID 25469685
- [Background] Nooyens AC, Baan CA, Spijkerman AM, Verschuren WM. Type 2 diabetes and cognitive decline in middle-aged men and women: the Doetinchem Cohort Study. Diabetes Care. 2010 Sep;33(9):1964-9. doi: 10.2337/dc09-2038. Epub 2010 Jun 2. PMID 20519662
- [Background] Spauwen PJ, Kohler S, Verhey FR, Stehouwer CD, van Boxtel MP. Effects of type 2 diabetes on 12-year cognitive change: results from the Maastricht Aging Study. Diabetes Care. 2013 Jun;36(6):1554-61. doi: 10.2337/dc12-0746. Epub 2012 Dec 28. PMID 23275366
- [Background] Worrall G, Moulton N, Briffett E. Effect of type II diabetes mellitus on cognitive function. J Fam Pract. 1993 Jun;36(6):639-43. PMID 8505607
- [Background] Lowe LP, Tranel D, Wallace RB, Welty TK. Type II diabetes and cognitive function. A population-based study of Native Americans. Diabetes Care. 1994 Aug;17(8):891-6. doi: 10.2337/diacare.17.8.891. PMID 7956638
- [Background] Dey J, Misra A, Desai NG, Mahapatra AK, Padma MV. Cognitive function in younger type II diabetes. Diabetes Care. 1997 Jan;20(1):32-5. doi: 10.2337/diacare.20.1.32. PMID 9028690
- [Background] McGuire LC, Ford ES, Ajani UA. The impact of cognitive functioning on mortality and the development of functional disability in older adults with diabetes: the second longitudinal study on aging. BMC Geriatr. 2006 May 1;6:8. doi: 10.1186/1471-2318-6-8. PMID 16650284
- [Background] Diaz-Venegas C, Schneider DC, Myrskyla M, Mehta NK. Life expectancy with and without cognitive impairment by diabetes status among older Americans. PLoS One. 2017 Dec 29;12(12):e0190488. doi: 10.1371/journal.pone.0190488. eCollection 2017. PMID 29287106
- [Background] Cuevas H, Stuifbergen A. Perceived cognitive deficits are associated with diabetes self-management in a multiethnic sample. J Diabetes Metab Disord. 2017 Feb 15;16:7. doi: 10.1186/s40200-017-0289-3. eCollection 2017. PMID 28239597
- [Background] Yaffe K, Lindquist K, Vittinghoff E, Barnes D, Simonsick EM, Newman A, Satterfield S, Rosano C, Rubin SM, Ayonayon HN, Harris T; Health, Aging and Body Compsition Study. The effect of maintaining cognition on risk of disability and death. J Am Geriatr Soc. 2010 May;58(5):889-94. doi: 10.1111/j.1532-5415.2010.02818.x. Epub 2010 Apr 6. PMID 20406308
- [Background] Lavery LL, Dodge HH, Snitz B, Ganguli M. Cognitive decline and mortality in a community-based cohort: the Monongahela Valley Independent Elders Survey. J Am Geriatr Soc. 2009 Jan;57(1):94-100. doi: 10.1111/j.1532-5415.2008.02052.x. Epub 2008 Nov 3. PMID 19016932
- [Background] Gatlin PK, Insel KC. Severity of Type 2 Diabetes, Cognitive Function, and Self-Care. Biol Res Nurs. 2015 Oct;17(5):540-8. doi: 10.1177/1099800414557565. Epub 2014 Nov 11. PMID 25391255
- [Background] Feil DG, Zhu CW, Sultzer DL. The relationship between cognitive impairment and diabetes self-management in a population-based community sample of older adults with Type 2 diabetes. J Behav Med. 2012 Apr;35(2):190-9. doi: 10.1007/s10865-011-9344-6. Epub 2011 Apr 19. PMID 21503710
- [Background] Tomlin A, Sinclair A. The influence of cognition on self-management of type 2 diabetes in older people. Psychol Res Behav Manag. 2016 Jan 21;9:7-20. doi: 10.2147/PRBM.S36238. eCollection 2016. PMID 26855601
- [Background] Rosen MI, Beauvais JE, Rigsby MO, Salahi JT, Ryan CE, Cramer JA. Neuropsychological correlates of suboptimal adherence to metformin. J Behav Med. 2003 Aug;26(4):349-60. doi: 10.1023/a:1024257027839. PMID 12921008
- [Background] Kazlauskaite R, Soni S, Evans AT, Graham K, Fisher B. Accuracy of self-monitored blood glucose in type 2 diabetes. Diabetes Technol Ther. 2009 Jun;11(6):385-92. doi: 10.1089/dia.2008.0111. PMID 19459768
- [Background] de Wet H, Levitt N, Tipping B. Executive cognitive impairment detected by simple bedside testing is associated with poor glycaemic control in type 2 diabetes. S Afr Med J. 2007 Nov;97(11):1074-6. PMID 18250916
- [Background] Okura T, Heisler M, Langa KM. Association between cognitive function and social support with glycemic control in adults with diabetes mellitus. J Am Geriatr Soc. 2009 Oct;57(10):1816-24. doi: 10.1111/j.1532-5415.2009.02431.x. Epub 2009 Aug 13. PMID 19682129
- [Background] Norris SL, Lau J, Smith SJ, Schmid CH, Engelgau MM. Self-management education for adults with type 2 diabetes: a meta-analysis of the effect on glycemic control. Diabetes Care. 2002 Jul;25(7):1159-71. doi: 10.2337/diacare.25.7.1159. PMID 12087014
- [Background] Norris SL, Engelgau MM, Narayan KM. Effectiveness of self-management training in type 2 diabetes: a systematic review of randomized controlled trials. Diabetes Care. 2001 Mar;24(3):561-87. doi: 10.2337/diacare.24.3.561. PMID 11289485
- [Background] Xu WL, von Strauss E, Qiu CX, Winblad B, Fratiglioni L. Uncontrolled diabetes increases the risk of Alzheimer's disease: a population-based cohort study. Diabetologia. 2009 Jun;52(6):1031-9. doi: 10.1007/s00125-009-1323-x. Epub 2009 Mar 12. PMID 19280172
- [Background] Vagelatos NT, Eslick GD. Type 2 diabetes as a risk factor for Alzheimer's disease: the confounders, interactions, and neuropathology associated with this relationship. Epidemiol Rev. 2013;35:152-60. doi: 10.1093/epirev/mxs012. Epub 2013 Jan 11. PMID 23314404
- [Background] Jayaraman A, Pike CJ. Alzheimer's disease and type 2 diabetes: multiple mechanisms contribute to interactions. Curr Diab Rep. 2014 Apr;14(4):476. doi: 10.1007/s11892-014-0476-2. PMID 24526623
- [Background] Brundel M, van den Heuvel M, de Bresser J, Kappelle LJ, Biessels GJ; Utrecht Diabetic Encephalopathy Study Group. Cerebral cortical thickness in patients with type 2 diabetes. J Neurol Sci. 2010 Dec 15;299(1-2):126-30. doi: 10.1016/j.jns.2010.08.048. PMID 20869085
- [Background] den Heijer T, Vermeer SE, van Dijk EJ, Prins ND, Koudstaal PJ, Hofman A, Breteler MM. Type 2 diabetes and atrophy of medial temporal lobe structures on brain MRI. Diabetologia. 2003 Dec;46(12):1604-10. doi: 10.1007/s00125-003-1235-0. Epub 2003 Nov 1. PMID 14595538
- [Background] Manschot SM, Biessels GJ, de Valk H, Algra A, Rutten GE, van der Grond J, Kappelle LJ; Utrecht Diabetic Encephalopathy Study Group. Metabolic and vascular determinants of impaired cognitive performance and abnormalities on brain magnetic resonance imaging in patients with type 2 diabetes. Diabetologia. 2007 Nov;50(11):2388-97. doi: 10.1007/s00125-007-0792-z. Epub 2007 Sep 2. PMID 17764005
- [Background] Moran C, Phan TG, Chen J, Blizzard L, Beare R, Venn A, Munch G, Wood AG, Forbes J, Greenaway TM, Pearson S, Srikanth V. Brain atrophy in type 2 diabetes: regional distribution and influence on cognition. Diabetes Care. 2013 Dec;36(12):4036-42. doi: 10.2337/dc13-0143. Epub 2013 Aug 12. PMID 23939539
- [Background] Reijmer YD, Brundel M, de Bresser J, Kappelle LJ, Leemans A, Biessels GJ; Utrecht Vascular Cognitive Impairment Study Group. Microstructural white matter abnormalities and cognitive functioning in type 2 diabetes: a diffusion tensor imaging study. Diabetes Care. 2013 Jan;36(1):137-44. doi: 10.2337/dc12-0493. Epub 2012 Sep 6. PMID 22961577
- [Background] Whitlow CT, Sink KM, Divers J, Smith SC, Xu J, Palmer ND, Hugenschmidt CE, Williamson JD, Bowden DW, Freedman BI, Maldjian JA. Effects of Type 2 Diabetes on Brain Structure and Cognitive Function: African American-Diabetes Heart Study MIND. AJNR Am J Neuroradiol. 2015 Sep;36(9):1648-53. doi: 10.3174/ajnr.A4321. Epub 2015 Jul 23. PMID 26206811
- [Background] Bokura H, Robinson RG. Long-term cognitive impairment associated with caudate stroke. Stroke. 1997 May;28(5):970-5. doi: 10.1161/01.str.28.5.970. PMID 9158635
- [Background] Chang LJ, Yarkoni T, Khaw MW, Sanfey AG. Decoding the role of the insula in human cognition: functional parcellation and large-scale reverse inference. Cereb Cortex. 2013 Mar;23(3):739-49. doi: 10.1093/cercor/bhs065. Epub 2012 Mar 20. PMID 22437053
- [Background] di Pellegrino G, Ciaramelli E, Ladavas E. The regulation of cognitive control following rostral anterior cingulate cortex lesion in humans. J Cogn Neurosci. 2007 Feb;19(2):275-86. doi: 10.1162/jocn.2007.19.2.275. PMID 17280516
- [Background] Gu X, Liu X, Van Dam NT, Hof PR, Fan J. Cognition-emotion integration in the anterior insular cortex. Cereb Cortex. 2013 Jan;23(1):20-7. doi: 10.1093/cercor/bhr367. Epub 2012 Jan 23. PMID 22275476
- [Background] Hahn B, Ross TJ, Stein EA. Cingulate activation increases dynamically with response speed under stimulus unpredictability. Cereb Cortex. 2007 Jul;17(7):1664-71. doi: 10.1093/cercor/bhl075. Epub 2006 Sep 8. PMID 16963517
- [Background] Hampson M, Driesen NR, Skudlarski P, Gore JC, Constable RT. Brain connectivity related to working memory performance. J Neurosci. 2006 Dec 20;26(51):13338-43. doi: 10.1523/JNEUROSCI.3408-06.2006. PMID 17182784
- [Background] Jiang J, Beck J, Heller K, Egner T. An insula-frontostriatal network mediates flexible cognitive control by adaptively predicting changing control demands. Nat Commun. 2015 Sep 22;6:8165. doi: 10.1038/ncomms9165. PMID 26391305
- [Background] Kelly C, Toro R, Di Martino A, Cox CL, Bellec P, Castellanos FX, Milham MP. A convergent functional architecture of the insula emerges across imaging modalities. Neuroimage. 2012 Jul 16;61(4):1129-42. doi: 10.1016/j.neuroimage.2012.03.021. Epub 2012 Mar 13. PMID 22440648
- [Background] Kumaran D, Maguire EA. The human hippocampus: cognitive maps or relational memory? J Neurosci. 2005 Aug 3;25(31):7254-9. doi: 10.1523/JNEUROSCI.1103-05.2005. PMID 16079407
- [Background] Leech R, Kamourieh S, Beckmann CF, Sharp DJ. Fractionating the default mode network: distinct contributions of the ventral and dorsal posterior cingulate cortex to cognitive control. J Neurosci. 2011 Mar 2;31(9):3217-24. doi: 10.1523/JNEUROSCI.5626-10.2011. PMID 21368033
- [Background] Manes F, Springer J, Jorge R, Robinson RG. Verbal memory impairment after left insular cortex infarction. J Neurol Neurosurg Psychiatry. 1999 Oct;67(4):532-4. doi: 10.1136/jnnp.67.4.532. PMID 10486407
- [Background] Nelson SM, Dosenbach NU, Cohen AL, Wheeler ME, Schlaggar BL, Petersen SE. Role of the anterior insula in task-level control and focal attention. Brain Struct Funct. 2010 Jun;214(5-6):669-80. doi: 10.1007/s00429-010-0260-2. Epub 2010 May 29. PMID 20512372
- [Background] SCOVILLE WB, MILNER B. Loss of recent memory after bilateral hippocampal lesions. J Neurol Neurosurg Psychiatry. 1957 Feb;20(1):11-21. doi: 10.1136/jnnp.20.1.11. No abstract available. PMID 13406589
- [Background] Seger CA, Cincotta CM. The roles of the caudate nucleus in human classification learning. J Neurosci. 2005 Mar 16;25(11):2941-51. doi: 10.1523/JNEUROSCI.3401-04.2005. PMID 15772354
- [Background] Squire LR. Memory and the hippocampus: a synthesis from findings with rats, monkeys, and humans. Psychol Rev. 1992 Apr;99(2):195-231. doi: 10.1037/0033-295x.99.2.195. PMID 1594723
- [Background] Desmond JE, Gabrieli JD, Glover GH. Dissociation of frontal and cerebellar activity in a cognitive task: evidence for a distinction between selection and search. Neuroimage. 1998 May;7(4 Pt 1):368-76. doi: 10.1006/nimg.1998.0340. PMID 9626676
- [Background] Eichenbaum H. Hippocampus: cognitive processes and neural representations that underlie declarative memory. Neuron. 2004 Sep 30;44(1):109-20. doi: 10.1016/j.neuron.2004.08.028. PMID 15450164
- [Background] Frith C, Dolan R. The role of the prefrontal cortex in higher cognitive functions. Brain Res Cogn Brain Res. 1996 Dec;5(1-2):175-81. doi: 10.1016/s0926-6410(96)00054-7. PMID 9049084
- [Background] Goto K, Hoshi Y, Sata M, Kawahara M, Takahashi M, Murohashi H. Role of the prefrontal cortex in the cognitive control of reaching movements: near-infrared spectroscopy study. J Biomed Opt. 2011 Dec;16(12):127003. doi: 10.1117/1.3658757. PMID 22191933
- [Background] Grafman J, Litvan I, Massaquoi S, Stewart M, Sirigu A, Hallett M. Cognitive planning deficit in patients with cerebellar atrophy. Neurology. 1992 Aug;42(8):1493-6. doi: 10.1212/wnl.42.8.1493. PMID 1641142
- [Background] Koechlin E, Basso G, Pietrini P, Panzer S, Grafman J. The role of the anterior prefrontal cortex in human cognition. Nature. 1999 May 13;399(6732):148-51. doi: 10.1038/20178. PMID 10335843
- [Background] Ravizza SM, McCormick CA, Schlerf JE, Justus T, Ivry RB, Fiez JA. Cerebellar damage produces selective deficits in verbal working memory. Brain. 2006 Feb;129(Pt 2):306-20. doi: 10.1093/brain/awh685. Epub 2005 Nov 29. PMID 16317024
- [Background] Rice K, Viscomi B, Riggins T, Redcay E. Amygdala volume linked to individual differences in mental state inference in early childhood and adulthood. Dev Cogn Neurosci. 2014 Apr;8:153-63. doi: 10.1016/j.dcn.2013.09.003. Epub 2013 Sep 26. PMID 24139023
- [Background] Rougier NP, Noelle DC, Braver TS, Cohen JD, O'Reilly RC. Prefrontal cortex and flexible cognitive control: rules without symbols. Proc Natl Acad Sci U S A. 2005 May 17;102(20):7338-43. doi: 10.1073/pnas.0502455102. Epub 2005 May 9. PMID 15883365
- [Background] Rubin RD, Watson PD, Duff MC, Cohen NJ. The role of the hippocampus in flexible cognition and social behavior. Front Hum Neurosci. 2014 Sep 30;8:742. doi: 10.3389/fnhum.2014.00742. eCollection 2014. PMID 25324753
- [Background] Schaefer A, Gray JR. A role for the human amygdala in higher cognition. Rev Neurosci. 2007;18(5):355-63. doi: 10.1515/revneuro.2007.18.5.355. PMID 19544622
- [Background] Schmahmann JD. Disorders of the cerebellum: ataxia, dysmetria of thought, and the cerebellar cognitive affective syndrome. J Neuropsychiatry Clin Neurosci. 2004 Summer;16(3):367-78. doi: 10.1176/jnp.16.3.367. PMID 15377747
- [Background] Schmahmann JD, Sherman JC. The cerebellar cognitive affective syndrome. Brain. 1998 Apr;121 ( Pt 4):561-79. doi: 10.1093/brain/121.4.561. PMID 9577385
- [Background] Stoodley CJ. The cerebellum and cognition: evidence from functional imaging studies. Cerebellum. 2012 Jun;11(2):352-65. doi: 10.1007/s12311-011-0260-7. PMID 21373864
- [Background] Stoodley CJ, Schmahmann JD. The cerebellum and language: evidence from patients with cerebellar degeneration. Brain Lang. 2009 Sep;110(3):149-53. doi: 10.1016/j.bandl.2009.07.006. Epub 2009 Aug 6. PMID 19664816
- [Background] Sweatt JD. Hippocampal function in cognition. Psychopharmacology (Berl). 2004 Jun;174(1):99-110. doi: 10.1007/s00213-004-1795-9. Epub 2004 Mar 2. PMID 15205881
- [Background] Joo EY, Tae WS, Lee MJ, Kang JW, Park HS, Lee JY, Suh M, Hong SB. Reduced brain gray matter concentration in patients with obstructive sleep apnea syndrome. Sleep. 2010 Feb;33(2):235-41. doi: 10.1093/sleep/33.2.235. PMID 20175407
- [Background] Kumar R, Chavez AS, Macey PM, Woo MA, Yan-Go FL, Harper RM. Altered global and regional brain mean diffusivity in patients with obstructive sleep apnea. J Neurosci Res. 2012 Oct;90(10):2043-52. doi: 10.1002/jnr.23083. Epub 2012 Jun 20. PMID 22715089
- [Background] Macey PM, Henderson LA, Macey KE, Alger JR, Frysinger RC, Woo MA, Harper RK, Yan-Go FL, Harper RM. Brain morphology associated with obstructive sleep apnea. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1382-7. doi: 10.1164/rccm.200201-050OC. PMID 12421746
- [Background] Macey PM, Kumar R, Woo MA, Valladares EM, Yan-Go FL, Harper RM. Brain structural changes in obstructive sleep apnea. Sleep. 2008 Jul;31(7):967-77. PMID 18652092
- [Background] Tummala S, Roy B, Vig R, Park B, Kang DW, Woo MA, Aysola R, Harper RM, Kumar R. Non-Gaussian Diffusion Imaging Shows Brain Myelin and Axonal Changes in Obstructive Sleep Apnea. J Comput Assist Tomogr. 2017 Mar/Apr;41(2):181-189. doi: 10.1097/RCT.0000000000000537. PMID 27801694
- [Background] Tummala S, Roy B, Park B, Kang DW, Woo MA, Harper RM, Kumar R. Associations between brain white matter integrity and disease severity in obstructive sleep apnea. J Neurosci Res. 2016 Oct;94(10):915-923. doi: 10.1002/jnr.23788. Epub 2016 Jun 18. PMID 27315771
- [Background] Tummala S, Palomares J, Kang DW, Park B, Woo MA, Harper RM, Kumar R. Global and Regional Brain Non-Gaussian Diffusion Changes in Newly Diagnosed Patients with Obstructive Sleep Apnea. Sleep. 2016 Jan 1;39(1):51-7. doi: 10.5665/sleep.5316. PMID 26285005
- [Background] Cross RL, Kumar R, Macey PM, Doering LV, Alger JR, Yan-Go FL, Harper RM. Neural alterations and depressive symptoms in obstructive sleep apnea patients. Sleep. 2008 Aug;31(8):1103-9. PMID 18714782
- [Background] Kumar R, Birrer BV, Macey PM, Woo MA, Gupta RK, Yan-Go FL, Harper RM. Reduced mammillary body volume in patients with obstructive sleep apnea. Neurosci Lett. 2008 Jun 27;438(3):330-4. doi: 10.1016/j.neulet.2008.04.071. Epub 2008 Apr 25. PMID 18486338
- [Background] Kumar R, Pham TT, Macey PM, Woo MA, Yan-Go FL, Harper RM. Abnormal myelin and axonal integrity in recently diagnosed patients with obstructive sleep apnea. Sleep. 2014 Apr 1;37(4):723-32. doi: 10.5665/sleep.3578. PMID 24899761
- [Background] Sasongko L, Link JM, Muzi M, Mankoff DA, Yang X, Collier AC, Shoner SC, Unadkat JD. Imaging P-glycoprotein transport activity at the human blood-brain barrier with positron emission tomography. Clin Pharmacol Ther. 2005 Jun;77(6):503-14. doi: 10.1016/j.clpt.2005.01.022. PMID 15961982
- [Background] Hara T, Iio M, Tsukiyama T, Yokoi F. Measurement of human blood brain barrier integrity using 11C-inulin and positron emission tomography. Eur J Nucl Med. 1988;14(4):173-6. doi: 10.1007/BF00257322. PMID 3262514
- [Background] Schlageter NL, Carson RE, Rapoport SI. Examination of blood-brain barrier permeability in dementia of the Alzheimer type with [68Ga]EDTA and positron emission tomography. J Cereb Blood Flow Metab. 1987 Feb;7(1):1-8. doi: 10.1038/jcbfm.1987.1. PMID 3100543
- [Background] Nyakale NE, Clauss RP, Nel HW, Sathekge MM. Blood-brain barrier integrity in a zolpidem-responder patient. S Afr Med J. 2012 Jul 31;102(10):790-1. doi: 10.7196/samj.5993. PMID 23034205
- [Background] Lorberboym M, Lampl Y, Sadeh M. Correlation of 99mTc-DTPA SPECT of the blood-brain barrier with neurologic outcome after acute stroke. J Nucl Med. 2003 Dec;44(12):1898-904. PMID 14660714
- [Background] Gilad R, Lampl Y, Eilam A, Boaz M, Loyberboim M. SPECT-DTPA as a tool for evaluating the blood-brain barrier in post-stroke seizures. J Neurol. 2012 Oct;259(10):2041-4. doi: 10.1007/s00415-012-6445-2. Epub 2012 Feb 10. PMID 22323212
- [Background] Armitage PA, Farrall AJ, Carpenter TK, Doubal FN, Wardlaw JM. Use of dynamic contrast-enhanced MRI to measure subtle blood-brain barrier abnormalities. Magn Reson Imaging. 2011 Apr;29(3):305-14. doi: 10.1016/j.mri.2010.09.002. Epub 2010 Oct 27. PMID 21030178
- [Background] Bergamino M, Saitta L, Barletta L, Bonzano L, Mancardi GL, Castellan L, Ravetti JL, Roccatagliata L. Measurement of blood-brain barrier permeability with t1-weighted dynamic contrast-enhanced MRI in brain tumors: a comparative study with two different algorithms. ISRN Neurosci. 2013 Feb 20;2013:905279. doi: 10.1155/2013/905279. eCollection 2013. PMID 24959569
- [Background] Larsson HB, Courivaud F, Rostrup E, Hansen AE. Measurement of brain perfusion, blood volume, and blood-brain barrier permeability, using dynamic contrast-enhanced T(1)-weighted MRI at 3 tesla. Magn Reson Med. 2009 Nov;62(5):1270-81. doi: 10.1002/mrm.22136. PMID 19780145
- [Background] Veksler R, Shelef I, Friedman A. Blood-brain barrier imaging in human neuropathologies. Arch Med Res. 2014 Nov;45(8):646-52. doi: 10.1016/j.arcmed.2014.11.016. Epub 2014 Nov 29. PMID 25453223
- [Background] Gotthardt M, Bleeker-Rovers CP, Boerman OC, Oyen WJ. Imaging of inflammation by PET, conventional scintigraphy, and other imaging techniques. J Nucl Med. 2010 Dec;51(12):1937-49. doi: 10.2967/jnumed.110.076232. Epub 2010 Nov 15. PMID 21078798
- [Background] Perazella MA. Gadolinium-contrast toxicity in patients with kidney disease: nephrotoxicity and nephrogenic systemic fibrosis. Curr Drug Saf. 2008 Jan;3(1):67-75. doi: 10.2174/157488608783333989. PMID 18690983
- [Background] Wang J, Fernandez-Seara MA, Wang S, St Lawrence KS. When perfusion meets diffusion: in vivo measurement of water permeability in human brain. J Cereb Blood Flow Metab. 2007 Apr;27(4):839-49. doi: 10.1038/sj.jcbfm.9600398. Epub 2006 Sep 13. PMID 16969383
- [Background] St Lawrence KS, Owen D, Wang DJ. A two-stage approach for measuring vascular water exchange and arterial transit time by diffusion-weighted perfusion MRI. Magn Reson Med. 2012 May;67(5):1275-84. doi: 10.1002/mrm.23104. Epub 2011 Aug 19. PMID 21858870
- [Background] Wang J, Alsop DC, Song HK, Maldjian JA, Tang K, Salvucci AE, Detre JA. Arterial transit time imaging with flow encoding arterial spin tagging (FEAST). Magn Reson Med. 2003 Sep;50(3):599-607. doi: 10.1002/mrm.10559. PMID 12939768
- [Background] Silva AC, Williams DS, Koretsky AP. Evidence for the exchange of arterial spin-labeled water with tissue water in rat brain from diffusion-sensitized measurements of perfusion. Magn Reson Med. 1997 Aug;38(2):232-7. doi: 10.1002/mrm.1910380211. PMID 9256102
- [Background] Tiwari YV, Lu J, Shen Q, Cerqueira B, Duong TQ. Magnetic resonance imaging of blood-brain barrier permeability in ischemic stroke using diffusion-weighted arterial spin labeling in rats. J Cereb Blood Flow Metab. 2017 Aug;37(8):2706-2715. doi: 10.1177/0271678X16673385. Epub 2016 Jan 1. PMID 27742887
- [Background] Peng L, Xu L, Ouyang W. Role of peripheral inflammatory markers in postoperative cognitive dysfunction (POCD): a meta-analysis. PLoS One. 2013 Nov 13;8(11):e79624. doi: 10.1371/journal.pone.0079624. eCollection 2013. PMID 24236147
- [Background] Ali MS, Harmer M, Vaughan R. Serum S100 protein as a marker of cerebral damage during cardiac surgery. Br J Anaesth. 2000 Aug;85(2):287-98. doi: 10.1093/bja/85.2.287. PMID 10992840
- [Background] Linstedt U, Meyer O, Kropp P, Berkau A, Tapp E, Zenz M. Serum concentration of S-100 protein in assessment of cognitive dysfunction after general anesthesia in different types of surgery. Acta Anaesthesiol Scand. 2002 Apr;46(4):384-9. doi: 10.1034/j.1399-6576.2002.460409.x. PMID 11952437
- [Background] Cao XZ, Ma H, Wang JK, Liu F, Wu BY, Tian AY, Wang LL, Tan WF. Postoperative cognitive deficits and neuroinflammation in the hippocampus triggered by surgical trauma are exacerbated in aged rats. Prog Neuropsychopharmacol Biol Psychiatry. 2010 Dec 1;34(8):1426-32. doi: 10.1016/j.pnpbp.2010.07.027. Epub 2010 Aug 4. PMID 20691747
- [Background] Chen J, Cui X, Zacharek A, Chopp M. Increasing Ang1/Tie2 expression by simvastatin treatment induces vascular stabilization and neuroblast migration after stroke. J Cell Mol Med. 2009 Jul;13(7):1348-57. doi: 10.1111/j.1582-4934.2008.00380.x. Epub 2008 Jun 9. PMID 18544044
- [Background] Ifergan I, Wosik K, Cayrol R, Kebir H, Auger C, Bernard M, Bouthillier A, Moumdjian R, Duquette P, Prat A. Statins reduce human blood-brain barrier permeability and restrict leukocyte migration: relevance to multiple sclerosis. Ann Neurol. 2006 Jul;60(1):45-55. doi: 10.1002/ana.20875. PMID 16729291
- [Background] Jiang JY, Lyeth BG, Kapasi MZ, Jenkins LW, Povlishock JT. Moderate hypothermia reduces blood-brain barrier disruption following traumatic brain injury in the rat. Acta Neuropathol. 1992;84(5):495-500. doi: 10.1007/BF00304468. PMID 1462764
- [Background] Miller DH, Thompson AJ, Morrissey SP, MacManus DG, Moore SG, Kendall BE, Moseley IF, McDonald WI. High dose steroids in acute relapses of multiple sclerosis: MRI evidence for a possible mechanism of therapeutic effect. J Neurol Neurosurg Psychiatry. 1992 Jun;55(6):450-3. doi: 10.1136/jnnp.55.6.450. PMID 1619410
- [Background] Yang D, Knight RA, Han Y, Karki K, Zhang J, Ding C, Chopp M, Seyfried DM. Vascular recovery promoted by atorvastatin and simvastatin after experimental intracerebral hemorrhage: magnetic resonance imaging and histological study. J Neurosurg. 2011 Apr;114(4):1135-42. doi: 10.3171/2010.7.JNS10163. Epub 2010 Aug 20. PMID 20722611
- [Background] Ahishali B, Kaya M, Orhan N, Arican N, Ekizoglu O, Elmas I, Kucuk M, Kemikler G, Kalayci R, Gurses C. Effects of levetiracetam on blood-brain barrier disturbances following hyperthermia-induced seizures in rats with cortical dysplasia. Life Sci. 2010 Nov 20;87(19-22):609-19. doi: 10.1016/j.lfs.2010.09.014. Epub 2010 Sep 25. PMID 20875430
- [Background] Chen X, Gawryluk JW, Wagener JF, Ghribi O, Geiger JD. Caffeine blocks disruption of blood brain barrier in a rabbit model of Alzheimer's disease. J Neuroinflammation. 2008 Apr 3;5:12. doi: 10.1186/1742-2094-5-12. PMID 18387175
- [Background] Gurses C, Orhan N, Ahishali B, Yilmaz CU, Kemikler G, Elmas I, Cevik A, Kucuk M, Arican N, Kaya M. Topiramate reduces blood-brain barrier disruption and inhibits seizure activity in hyperthermia-induced seizures in rats with cortical dysplasia. Brain Res. 2013 Feb 4;1494:91-100. doi: 10.1016/j.brainres.2012.11.039. Epub 2012 Nov 29. PMID 23201444
- [Background] Lehmann M, Regland B, Blennow K, Gottfries CG. Vitamin B12-B6-folate treatment improves blood-brain barrier function in patients with hyperhomocysteinaemia and mild cognitive impairment. Dement Geriatr Cogn Disord. 2003;16(3):145-50. doi: 10.1159/000071002. PMID 12826740
- [Background] Pfeiffer F, Schafer J, Lyck R, Makrides V, Brunner S, Schaeren-Wiemers N, Deutsch U, Engelhardt B. Claudin-1 induced sealing of blood-brain barrier tight junctions ameliorates chronic experimental autoimmune encephalomyelitis. Acta Neuropathol. 2011 Nov;122(5):601-14. doi: 10.1007/s00401-011-0883-2. Epub 2011 Oct 9. PMID 21983942
- [Background] Ueno Y, Zhang N, Miyamoto N, Tanaka R, Hattori N, Urabe T. Edaravone attenuates white matter lesions through endothelial protection in a rat chronic hypoperfusion model. Neuroscience. 2009 Aug 18;162(2):317-27. doi: 10.1016/j.neuroscience.2009.04.065. Epub 2009 May 3. PMID 19409967
- [Background] Schroth G, Wichmann W, Valavanis A. Blood-brain-barrier disruption in acute Wernicke encephalopathy: MR findings. J Comput Assist Tomogr. 1991 Nov-Dec;15(6):1059-61. doi: 10.1097/00004728-199111000-00034. PMID 1939760
- [Background] Arora S, Lidor A, Abularrage CJ, Weiswasser JM, Nylen E, Kellicut D, Sidawy AN. Thiamine (vitamin B1) improves endothelium-dependent vasodilatation in the presence of hyperglycemia. Ann Vasc Surg. 2006 Sep;20(5):653-8. doi: 10.1007/s10016-006-9055-6. Epub 2006 May 31. PMID 16741654
- [Background] Beltramo E, Berrone E, Buttiglieri S, Porta M. Thiamine and benfotiamine prevent increased apoptosis in endothelial cells and pericytes cultured in high glucose. Diabetes Metab Res Rev. 2004 Jul-Aug;20(4):330-6. doi: 10.1002/dmrr.470. PMID 15250036
- [Background] Stirban A, Pop A, Tschoepe D. A randomized, double-blind, crossover, placebo-controlled trial of 6 weeks benfotiamine treatment on postprandial vascular function and variables of autonomic nerve function in Type 2 diabetes. Diabet Med. 2013 Oct;30(10):1204-8. doi: 10.1111/dme.12240. Epub 2013 Jun 12. PMID 23701274
- [Background] Wong CY, Qiuwaxi J, Chen H, Li SW, Chan HT, Tam S, Shu XO, Lau CP, Kwong YL, Tse HF. Daily intake of thiamine correlates with the circulating level of endothelial progenitor cells and the endothelial function in patients with type II diabetes. Mol Nutr Food Res. 2008 Dec;52(12):1421-7. doi: 10.1002/mnfr.200800056. PMID 18925614
- [Background] Pomero F, Molinar Min A, La Selva M, Allione A, Molinatti GM, Porta M. Benfotiamine is similar to thiamine in correcting endothelial cell defects induced by high glucose. Acta Diabetol. 2001;38(3):135-8. doi: 10.1007/s005920170010. PMID 11827434
- [Background] Stirban A, Negrean M, Stratmann B, Gawlowski T, Horstmann T, Gotting C, Kleesiek K, Mueller-Roesel M, Koschinsky T, Uribarri J, Vlassara H, Tschoepe D. Benfotiamine prevents macro- and microvascular endothelial dysfunction and oxidative stress following a meal rich in advanced glycation end products in individuals with type 2 diabetes. Diabetes Care. 2006 Sep;29(9):2064-71. doi: 10.2337/dc06-0531. PMID 16936154
- [Background] Lonsdale D. A review of the biochemistry, metabolism and clinical benefits of thiamin(e) and its derivatives. Evid Based Complement Alternat Med. 2006 Mar;3(1):49-59. doi: 10.1093/ecam/nek009. PMID 16550223
- [Background] Kornreich L, Bron-Harlev E, Hoffmann C, Schwarz M, Konen O, Schoenfeld T, Straussberg R, Nahum E, Ibrahim AK, Eshel G, Horev G. Thiamine deficiency in infants: MR findings in the brain. AJNR Am J Neuroradiol. 2005 Aug;26(7):1668-74. PMID 16091511
- [Background] Harper C. Thiamine (vitamin B1) deficiency and associated brain damage is still common throughout the world and prevention is simple and safe! Eur J Neurol. 2006 Oct;13(10):1078-82. doi: 10.1111/j.1468-1331.2006.01530.x. PMID 16987159
- [Background] Calingasan NY, Chun WJ, Park LC, Uchida K, Gibson GE. Oxidative stress is associated with region-specific neuronal death during thiamine deficiency. J Neuropathol Exp Neurol. 1999 Sep;58(9):946-58. doi: 10.1097/00005072-199909000-00005. PMID 10499437
- [Background] Langlais PJ, Savage LM. Thiamine deficiency in rats produces cognitive and memory deficits on spatial tasks that correlate with tissue loss in diencephalon, cortex and white matter. Behav Brain Res. 1995 Apr;68(1):75-89. doi: 10.1016/0166-4328(94)00162-9. PMID 7619308
- [Background] Anwar A, Ahmed Azmi M, Siddiqui JA, Panhwar G, Shaikh F, Ariff M. Thiamine Level in Type I and Type II Diabetes Mellitus Patients: A Comparative Study Focusing on Hematological and Biochemical Evaluations. Cureus. 2020 May 8;12(5):e8027. doi: 10.7759/cureus.8027. PMID 32528766
- [Background] Jermendy G. Evaluating thiamine deficiency in patients with diabetes. Diab Vasc Dis Res. 2006 Sep;3(2):120-1. doi: 10.3132/dvdr.2006.014. No abstract available. PMID 17058632
- [Background] Thornalley PJ, Babaei-Jadidi R, Al Ali H, Rabbani N, Antonysunil A, Larkin J, Ahmed A, Rayman G, Bodmer CW. High prevalence of low plasma thiamine concentration in diabetes linked to a marker of vascular disease. Diabetologia. 2007 Oct;50(10):2164-70. doi: 10.1007/s00125-007-0771-4. Epub 2007 Aug 4. PMID 17676306
- [Background] Al-Attas OS, Al-Daghri NM, Alfadda AA, Abd-Alrahman SH, Sabico S. Blood thiamine and its phosphate esters as measured by high-performance liquid chromatography: levels and associations in diabetes mellitus patients with varying degrees of microalbuminuria. J Endocrinol Invest. 2012 Dec;35(11):951-6. doi: 10.3275/8126. Epub 2011 Nov 22. PMID 22107884
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Smith T, Gildeh N, Holmes C. The Montreal Cognitive Assessment: validity and utility in a memory clinic setting. Can J Psychiatry. 2007 May;52(5):329-32. doi: 10.1177/070674370705200508. PMID 17542384
- [Background] Hameed I, Masoodi SR, Mir SA, Nabi M, Ghazanfar K, Ganai BA. Type 2 diabetes mellitus: From a metabolic disorder to an inflammatory condition. World J Diabetes. 2015 May 15;6(4):598-612. doi: 10.4239/wjd.v6.i4.598. PMID 25987957
- [Background] Daousi C, Casson IF, Gill GV, MacFarlane IA, Wilding JP, Pinkney JH. Prevalence of obesity in type 2 diabetes in secondary care: association with cardiovascular risk factors. Postgrad Med J. 2006 Apr;82(966):280-4. doi: 10.1136/pmj.2005.039032. PMID 16597817
- [Background] Fletcher B, Gulanick M, Lamendola C. Risk factors for type 2 diabetes mellitus. J Cardiovasc Nurs. 2002 Jan;16(2):17-23. doi: 10.1097/00005082-200201000-00003. PMID 11800065
- [Background] Boyle JP, Thompson TJ, Gregg EW, Barker LE, Williamson DF. Projection of the year 2050 burden of diabetes in the US adult population: dynamic modeling of incidence, mortality, and prediabetes prevalence. Popul Health Metr. 2010 Oct 22;8:29. doi: 10.1186/1478-7954-8-29. PMID 20969750
- [Background] American Diabetes Association. Economic costs of diabetes in the U.S. in 2012. Diabetes Care. 2013 Apr;36(4):1033-46. doi: 10.2337/dc12-2625. Epub 2013 Mar 6. PMID 23468086
- [Background] van den Berg E, Reijmer YD, de Bresser J, Kessels RP, Kappelle LJ, Biessels GJ; Utrecht Diabetic Encephalopathy Study Group. A 4 year follow-up study of cognitive functioning in patients with type 2 diabetes mellitus. Diabetologia. 2010 Jan;53(1):58-65. doi: 10.1007/s00125-009-1571-9. Epub 2009 Oct 31. PMID 19882137
- [Background] Ebady SA, Arami MA, Shafigh MH. Investigation on the relationship between diabetes mellitus type 2 and cognitive impairment. Diabetes Res Clin Pract. 2008 Dec;82(3):305-9. doi: 10.1016/j.diabres.2008.08.020. Epub 2008 Oct 9. PMID 18848366
- [Background] Ruis C, Biessels GJ, Gorter KJ, van den Donk M, Kappelle LJ, Rutten GE. Cognition in the early stage of type 2 diabetes. Diabetes Care. 2009 Jul;32(7):1261-5. doi: 10.2337/dc08-2143. Epub 2009 Apr 14. PMID 19366968
- [Background] Yau PL, Kluger A, Borod JC, Convit A. Neural substrates of verbal memory impairments in adults with type 2 diabetes mellitus. J Clin Exp Neuropsychol. 2014;36(1):74-87. doi: 10.1080/13803395.2013.869310. Epub 2014 Jan 14. PMID 24417611
- [Background] Hassing LB, Grant MD, Hofer SM, Pedersen NL, Nilsson SE, Berg S, McClearn G, Johansson B. Type 2 diabetes mellitus contributes to cognitive decline in old age: a longitudinal population-based study. J Int Neuropsychol Soc. 2004 Jul;10(4):599-607. doi: 10.1017/S1355617704104165. PMID 15327738
- [Background] Arvanitakis Z, Wilson RS, Li Y, Aggarwal NT, Bennett DA. Diabetes and function in different cognitive systems in older individuals without dementia. Diabetes Care. 2006 Mar;29(3):560-5. doi: 10.2337/diacare.29.03.06.dc05-1901. PMID 16505506
- [Background] Fitas A, Orzechowska A, Juszczak D, Talarowska M. [Working memory in patients with type 2 diabetes]. Pol Merkur Lekarski. 2010 May;28(167):376-8. Polish. PMID 20568401
- [Background] Takeuchi A, Matsushima E, Kato M, Konishi M, Izumiyama H, Murata Y, Hirata Y. Characteristics of neuropsychological functions in inpatients with poorly-controlled type 2 diabetes mellitus. J Diabetes Investig. 2012 Jun 6;3(3):325-30. doi: 10.1111/j.2040-1124.2011.00170.x. PMID 24843583
- [Background] Mooradian AD, Perryman K, Fitten J, Kavonian GD, Morley JE. Cortical function in elderly non-insulin dependent diabetic patients. Behavioral and electrophysiologic studies. Arch Intern Med. 1988 Nov;148(11):2369-72. PMID 3190370
- [Background] Ryan CM, Geckle MO. Circumscribed cognitive dysfunction in middle-aged adults with type 2 diabetes. Diabetes Care. 2000 Oct;23(10):1486-93. doi: 10.2337/diacare.23.10.1486. PMID 11023141
- [Background] Schmitz N, Gariepy G, Smith KJ, Clyde M, Malla A, Boyer R, Strychar I, Lesage A, Wang J. Recurrent subthreshold depression in type 2 diabetes: an important risk factor for poor health outcomes. Diabetes Care. 2014 Apr;37(4):970-8. doi: 10.2337/dc13-1832. Epub 2013 Nov 6. PMID 24198303
- [Background] Monette MC, Baird A, Jackson DL. A meta-analysis of cognitive functioning in nondemented adults with type 2 diabetes mellitus. Can J Diabetes. 2014 Dec;38(6):401-8. doi: 10.1016/j.jcjd.2014.01.014. Epub 2014 Jun 3. PMID 24933107
- [Background] Manschot SM, Brands AM, van der Grond J, Kessels RP, Algra A, Kappelle LJ, Biessels GJ; Utrecht Diabetic Encephalopathy Study Group. Brain magnetic resonance imaging correlates of impaired cognition in patients with type 2 diabetes. Diabetes. 2006 Apr;55(4):1106-13. doi: 10.2337/diabetes.55.04.06.db05-1323. PMID 16567535
- [Background] Strachan MW, Deary IJ, Ewing FM, Frier BM. Is type II diabetes associated with an increased risk of cognitive dysfunction? A critical review of published studies. Diabetes Care. 1997 Mar;20(3):438-45. doi: 10.2337/diacare.20.3.438. PMID 9051402
- [Background] Ding J, Strachan MW, Reynolds RM, Frier BM, Deary IJ, Fowkes FG, Lee AJ, McKnight J, Halpin P, Swa K, Price JF; Edinburgh Type 2 Diabetes Study Investigators. Diabetic retinopathy and cognitive decline in older people with type 2 diabetes: the Edinburgh Type 2 Diabetes Study. Diabetes. 2010 Nov;59(11):2883-9. doi: 10.2337/db10-0752. Epub 2010 Aug 26. PMID 20798334
- [Background] Li C, Barker L, Ford ES, Zhang X, Strine TW, Mokdad AH. Diabetes and anxiety in US adults: findings from the 2006 Behavioral Risk Factor Surveillance System. Diabet Med. 2008 Jul;25(7):878-81. doi: 10.1111/j.1464-5491.2008.02477.x. PMID 18644077
- [Background] Li C, Ford ES, Strine TW, Mokdad AH. Prevalence of depression among U.S. adults with diabetes: findings from the 2006 behavioral risk factor surveillance system. Diabetes Care. 2008 Jan;31(1):105-7. doi: 10.2337/dc07-1154. Epub 2007 Oct 12. PMID 17934145
- [Background] Kent D, D'Eramo Melkus G, Stuart PM, McKoy JM, Urbanski P, Boren SA, Coke L, Winters JE, Horsley NL, Sherr D, Lipman R. Reducing the risks of diabetes complications through diabetes self-management education and support. Popul Health Manag. 2013 Apr;16(2):74-81. doi: 10.1089/pop.2012.0020. Epub 2013 Feb 13. PMID 23405872
- [Background] Mehravar F, Mansournia MA, Holakouie-Naieni K, Nasli-Esfahani E, Mansournia N, Almasi-Hashiani A. Associations between diabetes self-management and microvascular complications in patients with type 2 diabetes. Epidemiol Health. 2016 Jan 25;38:e2016004. doi: 10.4178/epih/e2016004. eCollection 2016. PMID 26883737
- [Background] Cui Y, Liang X, Gu H, Hu Y, Zhao Z, Yang XY, Qian C, Yang Y, Teng GJ. Cerebral perfusion alterations in type 2 diabetes and its relation to insulin resistance and cognitive dysfunction. Brain Imaging Behav. 2017 Oct;11(5):1248-1257. doi: 10.1007/s11682-016-9583-9. PMID 27714551
- [Background] Kumar A, Gupta R, Thomas A, Ajilore O, Hellemann G. Focal subcortical biophysical abnormalities in patients diagnosed with type 2 diabetes and depression. Arch Gen Psychiatry. 2009 Mar;66(3):324-30. doi: 10.1001/archgenpsychiatry.2008.548. PMID 19255382
- [Background] Starr JM, Wardlaw J, Ferguson K, MacLullich A, Deary IJ, Marshall I. Increased blood-brain barrier permeability in type II diabetes demonstrated by gadolinium magnetic resonance imaging. J Neurol Neurosurg Psychiatry. 2003 Jan;74(1):70-6. doi: 10.1136/jnnp.74.1.70. PMID 12486269
- [Background] Seaquist ER. The final frontier: how does diabetes affect the brain? Diabetes. 2010 Jan;59(1):4-5. doi: 10.2337/db09-1600. No abstract available. PMID 20040482
- [Background] Pugazhenthi S, Qin L, Reddy PH. Common neurodegenerative pathways in obesity, diabetes, and Alzheimer's disease. Biochim Biophys Acta Mol Basis Dis. 2017 May;1863(5):1037-1045. doi: 10.1016/j.bbadis.2016.04.017. Epub 2016 May 6. PMID 27156888
- [Background] Ryan JP, Fine DF, Rosano C. Type 2 diabetes and cognitive impairment: contributions from neuroimaging. J Geriatr Psychiatry Neurol. 2014 Mar;27(1):47-55. doi: 10.1177/0891988713516543. Epub 2014 Jan 5. PMID 24394151
- [Background] Roy B, Ehlert L, Mullur R, Freeby MJ, Woo MA, Kumar R, Choi S. Regional Brain Gray Matter Changes in Patients with Type 2 Diabetes Mellitus. Sci Rep. 2020 Jun 18;10(1):9925. doi: 10.1038/s41598-020-67022-5. PMID 32555374
- [Background] Geissler A, Frund R, Scholmerich J, Feuerbach S, Zietz B. Alterations of cerebral metabolism in patients with diabetes mellitus studied by proton magnetic resonance spectroscopy. Exp Clin Endocrinol Diabetes. 2003 Oct;111(7):421-7. doi: 10.1055/s-2003-44289. PMID 14614649
- [Background] Lin Y, Zhou J, Sha L, Li Y, Qu X, Liu L, Chen H, An Z, Wang Y, Sun C. Metabolite differences in the lenticular nucleus in type 2 diabetes mellitus shown by proton MR spectroscopy. AJNR Am J Neuroradiol. 2013 Sep;34(9):1692-6. doi: 10.3174/ajnr.A3492. Epub 2013 Apr 18. PMID 23598834
- [Background] Ajilore O, Haroon E, Kumaran S, Darwin C, Binesh N, Mintz J, Miller J, Thomas MA, Kumar A. Measurement of brain metabolites in patients with type 2 diabetes and major depression using proton magnetic resonance spectroscopy. Neuropsychopharmacology. 2007 Jun;32(6):1224-31. doi: 10.1038/sj.npp.1301248. Epub 2006 Dec 20. PMID 17180124
- [Background] Sahin I, Alkan A, Keskin L, Cikim A, Karakas HM, Firat AK, Sigirci A. Evaluation of in vivo cerebral metabolism on proton magnetic resonance spectroscopy in patients with impaired glucose tolerance and type 2 diabetes mellitus. J Diabetes Complications. 2008 Jul-Aug;22(4):254-60. doi: 10.1016/j.jdiacomp.2007.03.007. Epub 2008 Apr 16. PMID 18413166
- [Background] Kreis R, Ross BD. Cerebral metabolic disturbances in patients with subacute and chronic diabetes mellitus: detection with proton MR spectroscopy. Radiology. 1992 Jul;184(1):123-30. doi: 10.1148/radiology.184.1.1319074.
- [Background] Hsu JL, Chen YL, Leu JG, Jaw FS, Lee CH, Tsai YF, Hsu CY, Bai CH, Leemans A. Microstructural white matter abnormalities in type 2 diabetes mellitus: a diffusion tensor imaging study. Neuroimage. 2012 Jan 16;59(2):1098-105. doi: 10.1016/j.neuroimage.2011.09.041. Epub 2011 Sep 24. PMID 21967726
- [Background] Tan X, Fang P, An J, Lin H, Liang Y, Shen W, Leng X, Zhang C, Zheng Y, Qiu S. Micro-structural white matter abnormalities in type 2 diabetic patients: a DTI study using TBSS analysis. Neuroradiology. 2016 Dec;58(12):1209-1216. doi: 10.1007/s00234-016-1752-4. Epub 2016 Oct 25. PMID 27783100
- [Background] Yau PL, Javier D, Tsui W, Sweat V, Bruehl H, Borod JC, Convit A. Emotional and neutral declarative memory impairments and associated white matter microstructural abnormalities in adults with type 2 diabetes. Psychiatry Res. 2009 Dec 30;174(3):223-30. doi: 10.1016/j.pscychresns.2009.04.016. Epub 2009 Nov 10. PMID 19906514
- [Background] Zhang J, Wang Y, Wang J, Zhou X, Shu N, Wang Y, Zhang Z. White matter integrity disruptions associated with cognitive impairments in type 2 diabetic patients. Diabetes. 2014 Nov;63(11):3596-605. doi: 10.2337/db14-0342. Epub 2014 Jun 19. PMID 24947353
- [Background] Xiong Y, Sui Y, Xu Z, Zhang Q, Karaman MM, Cai K, Anderson TM, Zhu W, Wang J, Zhou XJ. A Diffusion Tensor Imaging Study on White Matter Abnormalities in Patients with Type 2 Diabetes Using Tract-Based Spatial Statistics. AJNR Am J Neuroradiol. 2016 Aug;37(8):1462-9. doi: 10.3174/ajnr.A4740. Epub 2016 Mar 17. PMID 26988810
- [Background] Shibata H. Topographic organization of subcortical projections to the anterior thalamic nuclei in the rat. J Comp Neurol. 1992 Sep 1;323(1):117-27. doi: 10.1002/cne.903230110. PMID 1385491
- [Background] Aggleton JP, Vann SD, Saunders RC. Projections from the hippocampal region to the mammillary bodies in macaque monkeys. Eur J Neurosci. 2005 Nov;22(10):2519-30. doi: 10.1111/j.1460-9568.2005.04450.x. PMID 16307594
- [Background] Aggleton JP, Brown MW. Episodic memory, amnesia, and the hippocampal-anterior thalamic axis. Behav Brain Sci. 1999 Jun;22(3):425-44; discussion 444-89. PMID 11301518
- [Background] Campbell S, Macqueen G. The role of the hippocampus in the pathophysiology of major depression. J Psychiatry Neurosci. 2004 Nov;29(6):417-26. PMID 15644983
- [Background] Liu W, Ge T, Leng Y, Pan Z, Fan J, Yang W, Cui R. The Role of Neural Plasticity in Depression: From Hippocampus to Prefrontal Cortex. Neural Plast. 2017;2017:6871089. doi: 10.1155/2017/6871089. Epub 2017 Jan 26. PMID 28246558
- [Background] Miller EK. The prefrontal cortex and cognitive control. Nat Rev Neurosci. 2000 Oct;1(1):59-65. doi: 10.1038/35036228. PMID 11252769
- [Background] Duncan J, Owen AM. Common regions of the human frontal lobe recruited by diverse cognitive demands. Trends Neurosci. 2000 Oct;23(10):475-83. doi: 10.1016/s0166-2236(00)01633-7. PMID 11006464
- [Background] MacDonald AW 3rd, Cohen JD, Stenger VA, Carter CS. Dissociating the role of the dorsolateral prefrontal and anterior cingulate cortex in cognitive control. Science. 2000 Jun 9;288(5472):1835-8. doi: 10.1126/science.288.5472.1835. PMID 10846167
- [Background] Pandya DN, Yeterian EH. Comparison of prefrontal architecture and connections. Philos Trans R Soc Lond B Biol Sci. 1996 Oct 29;351(1346):1423-32. doi: 10.1098/rstb.1996.0127. PMID 8941954
- [Background] Quintana J, Fuster JM. From perception to action: temporal integrative functions of prefrontal and parietal neurons. Cereb Cortex. 1999 Apr-May;9(3):213-21. doi: 10.1093/cercor/9.3.213. PMID 10355901
- [Background] Parent A. Extrinsic connections of the basal ganglia. Trends Neurosci. 1990 Jul;13(7):254-8. doi: 10.1016/0166-2236(90)90105-j. PMID 1695399
- [Background] Parent A, Hazrati LN. Functional anatomy of the basal ganglia. I. The cortico-basal ganglia-thalamo-cortical loop. Brain Res Brain Res Rev. 1995 Jan;20(1):91-127. doi: 10.1016/0165-0173(94)00007-c. PMID 7711769
- [Background] Bush G, Luu P, Posner MI. Cognitive and emotional influences in anterior cingulate cortex. Trends Cogn Sci. 2000 Jun;4(6):215-222. doi: 10.1016/s1364-6613(00)01483-2. PMID 10827444
- [Background] Ebert D, Ebmeier KP. The role of the cingulate gyrus in depression: from functional anatomy to neurochemistry. Biol Psychiatry. 1996 Jun 15;39(12):1044-50. doi: 10.1016/0006-3223(95)00320-7. PMID 8780840
- [Background] Drevets WC, Savitz J, Trimble M. The subgenual anterior cingulate cortex in mood disorders. CNS Spectr. 2008 Aug;13(8):663-81. doi: 10.1017/s1092852900013754. PMID 18704022
- [Background] Menon V, Uddin LQ. Saliency, switching, attention and control: a network model of insula function. Brain Struct Funct. 2010 Jun;214(5-6):655-67. doi: 10.1007/s00429-010-0262-0. Epub 2010 May 29. PMID 20512370
- [Background] Reynolds SM, Zahm DS. Specificity in the projections of prefrontal and insular cortex to ventral striatopallidum and the extended amygdala. J Neurosci. 2005 Dec 14;25(50):11757-67. doi: 10.1523/JNEUROSCI.3432-05.2005. PMID 16354934
- [Background] Paulus MP, Stein MB. Interoception in anxiety and depression. Brain Struct Funct. 2010 Jun;214(5-6):451-63. doi: 10.1007/s00429-010-0258-9. Epub 2010 May 21. PMID 20490545
- [Background] Gogolla N. The insular cortex. Curr Biol. 2017 Jun 19;27(12):R580-R586. doi: 10.1016/j.cub.2017.05.010. PMID 28633023
- [Background] Carmichael ST, Price JL. Limbic connections of the orbital and medial prefrontal cortex in macaque monkeys. J Comp Neurol. 1995 Dec 25;363(4):615-641. doi: 10.1002/cne.903630408. PMID 8847421
- [Background] Myers-Schulz B, Koenigs M. Functional anatomy of ventromedial prefrontal cortex: implications for mood and anxiety disorders. Mol Psychiatry. 2012 Feb;17(2):132-41. doi: 10.1038/mp.2011.88. Epub 2011 Jul 26. PMID 21788943
- [Background] Ducharme S, Albaugh MD, Hudziak JJ, Botteron KN, Nguyen TV, Truong C, Evans AC, Karama S; Brain Development Cooperative Group. Anxious/depressed symptoms are linked to right ventromedial prefrontal cortical thickness maturation in healthy children and young adults. Cereb Cortex. 2014 Nov;24(11):2941-50. doi: 10.1093/cercor/bht151. Epub 2013 Jun 7. PMID 23749874
- [Background] Drevets WC. Neuroimaging abnormalities in the amygdala in mood disorders. Ann N Y Acad Sci. 2003 Apr;985:420-44. doi: 10.1111/j.1749-6632.2003.tb07098.x. PMID 12724175
- [Background] Martin EI, Ressler KJ, Binder E, Nemeroff CB. The neurobiology of anxiety disorders: brain imaging, genetics, and psychoneuroendocrinology. Psychiatr Clin North Am. 2009 Sep;32(3):549-75. doi: 10.1016/j.psc.2009.05.004. PMID 19716990
- [Background] Shin LM, Liberzon I. The neurocircuitry of fear, stress, and anxiety disorders. Neuropsychopharmacology. 2010 Jan;35(1):169-91. doi: 10.1038/npp.2009.83. PMID 19625997
- [Background] Habas C, Kamdar N, Nguyen D, Prater K, Beckmann CF, Menon V, Greicius MD. Distinct cerebellar contributions to intrinsic connectivity networks. J Neurosci. 2009 Jul 1;29(26):8586-94. doi: 10.1523/JNEUROSCI.1868-09.2009. PMID 19571149
- [Background] Krienen FM, Buckner RL. Segregated fronto-cerebellar circuits revealed by intrinsic functional connectivity. Cereb Cortex. 2009 Oct;19(10):2485-97. doi: 10.1093/cercor/bhp135. Epub 2009 Jul 10. PMID 19592571
- [Background] D'Angelo E, Casali S. Seeking a unified framework for cerebellar function and dysfunction: from circuit operations to cognition. Front Neural Circuits. 2013 Jan 10;6:116. doi: 10.3389/fncir.2012.00116. eCollection 2012. PMID 23335884
- [Background] Sandoval KE, Witt KA. Blood-brain barrier tight junction permeability and ischemic stroke. Neurobiol Dis. 2008 Nov;32(2):200-19. doi: 10.1016/j.nbd.2008.08.005. Epub 2008 Aug 27. PMID 18790057
- [Background] Pop V, Sorensen DW, Kamper JE, Ajao DO, Murphy MP, Head E, Hartman RE, Badaut J. Early brain injury alters the blood-brain barrier phenotype in parallel with beta-amyloid and cognitive changes in adulthood. J Cereb Blood Flow Metab. 2013 Feb;33(2):205-14. doi: 10.1038/jcbfm.2012.154. Epub 2012 Nov 14. PMID 23149553
- [Background] Mayhan WG. Disruption of blood-brain barrier during acute hypertension in adult and aged rats. Am J Physiol. 1990 Jun;258(6 Pt 2):H1735-8. doi: 10.1152/ajpheart.1990.258.6.H1735. PMID 2113773
- [Background] McKean S. Induced moderate hypothermia after cardiac arrest. AACN Adv Crit Care. 2009 Oct-Dec;20(4):342-53; quiz 354-5. doi: 10.1097/NCI.0b013e3181bcea4e. PMID 19893373
- [Background] Ennis SR, Keep RF. Effect of sustained-mild and transient-severe hyperglycemia on ischemia-induced blood-brain barrier opening. J Cereb Blood Flow Metab. 2007 Sep;27(9):1573-82. doi: 10.1038/sj.jcbfm.9600454. Epub 2007 Feb 7. PMID 17293843
- [Background] Dietrich WD, Alonso O, Busto R. Moderate hyperglycemia worsens acute blood-brain barrier injury after forebrain ischemia in rats. Stroke. 1993 Jan;24(1):111-6. doi: 10.1161/01.str.24.1.111. PMID 8418533
- [Background] Kamada H, Yu F, Nito C, Chan PH. Influence of hyperglycemia on oxidative stress and matrix metalloproteinase-9 activation after focal cerebral ischemia/reperfusion in rats: relation to blood-brain barrier dysfunction. Stroke. 2007 Mar;38(3):1044-9. doi: 10.1161/01.STR.0000258041.75739.cb. Epub 2007 Feb 1. PMID 17272778
- [Background] Yoo DY, Yim HS, Jung HY, Nam SM, Kim JW, Choi JH, Seong JK, Yoon YS, Kim DW, Hwang IK. Chronic type 2 diabetes reduces the integrity of the blood-brain barrier by reducing tight junction proteins in the hippocampus. J Vet Med Sci. 2016 Jul 1;78(6):957-62. doi: 10.1292/jvms.15-0589. Epub 2016 Feb 15. PMID 26876499
- [Background] Cai L, Li W, Zeng R, Cao Z, Guo Q, Huang Q, Liu X. Valsartan alleviates the blood-brain barrier dysfunction in db/db diabetic mice. Bioengineered. 2021 Dec;12(1):9070-9080. doi: 10.1080/21655979.2021.1981799. PMID 34697992
- [Background] Lee JY, Park CS, Choi HY, Yune TY. Ginseng Extracts, GS-KG9 and GS-E3D, Prevent Blood-Brain Barrier Disruption and Thereby Inhibit Apoptotic Cell Death of Hippocampal Neurons in Streptozotocin-Induced Diabetic Rats. Nutrients. 2020 Aug 9;12(8):2383. doi: 10.3390/nu12082383. PMID 32784852
- [Background] Prasad S, Sajja RK, Naik P, Cucullo L. Diabetes Mellitus and Blood-Brain Barrier Dysfunction: An Overview. J Pharmacovigil. 2014 Jun;2(2):125. doi: 10.4172/2329-6887.1000125. PMID 25632404
- [Background] Serlin Y, Levy J, Shalev H. Vascular pathology and blood-brain barrier disruption in cognitive and psychiatric complications of type 2 diabetes mellitus. Cardiovasc Psychiatry Neurol. 2011;2011:609202. doi: 10.1155/2011/609202. Epub 2011 Feb 17. PMID 21350721
- [Background] Mooradian AD. Central nervous system complications of diabetes mellitus--a perspective from the blood-brain barrier. Brain Res Brain Res Rev. 1997 Apr;23(3):210-8. doi: 10.1016/s0165-0173(97)00003-9. PMID 9164671
- [Background] Rhea EM, Banks WA. Role of the Blood-Brain Barrier in Central Nervous System Insulin Resistance. Front Neurosci. 2019 Jun 4;13:521. doi: 10.3389/fnins.2019.00521. eCollection 2019. PMID 31213970
- [Background] van Sloten TT, Sedaghat S, Carnethon MR, Launer LJ, Stehouwer CDA. Cerebral microvascular complications of type 2 diabetes: stroke, cognitive dysfunction, and depression. Lancet Diabetes Endocrinol. 2020 Apr;8(4):325-336. doi: 10.1016/S2213-8587(19)30405-X. Epub 2020 Mar 2. PMID 32135131
- [Background] Dhir S, Tarasenko M, Napoli E, Giulivi C. Neurological, Psychiatric, and Biochemical Aspects of Thiamine Deficiency in Children and Adults. Front Psychiatry. 2019 Apr 4;10:207. doi: 10.3389/fpsyt.2019.00207. eCollection 2019. PMID 31019473
- [Background] Butterworth RF. Effects of thiamine deficiency on brain metabolism: implications for the pathogenesis of the Wernicke-Korsakoff syndrome. Alcohol Alcohol. 1989;24(4):271-9. doi: 10.1093/oxfordjournals.alcalc.a044913. PMID 2675860
- [Background] Sriram K, Manzanares W, Joseph K. Thiamine in nutrition therapy. Nutr Clin Pract. 2012 Feb;27(1):41-50. doi: 10.1177/0884533611426149. Epub 2012 Jan 4. PMID 22223666
- [Background] Attaluri P, Castillo A, Edriss H, Nugent K. Thiamine Deficiency: An Important Consideration in Critically Ill Patients. Am J Med Sci. 2018 Oct;356(4):382-390. doi: 10.1016/j.amjms.2018.06.015. Epub 2018 Jun 21. PMID 30146080
- [Background] Page GL, Laight D, Cummings MH. Thiamine deficiency in diabetes mellitus and the impact of thiamine replacement on glucose metabolism and vascular disease. Int J Clin Pract. 2011 Jun;65(6):684-90. doi: 10.1111/j.1742-1241.2011.02680.x. PMID 21564442
- [Background] Lomivorotov VV, Moroz G, Ismoilov S, Shmyrev V, Efremov S, Abubakirov M, Batalov V, Landoni G, Lembo R, Bogachev-Prokophiev A, Sapegin A, Bellomo R. Sustained High-dose Thiamine Supplementation in High-risk Cardiac Patients Undergoing Cardiopulmonary Bypass: A Pilot Feasibility Study (The APPLY trial). J Cardiothorac Vasc Anesth. 2020 Mar;34(3):594-600. doi: 10.1053/j.jvca.2019.08.044. Epub 2019 Sep 4. PMID 31558398
- [Background] Brady JA, Rock CL, Horneffer MR. Thiamin status, diuretic medications, and the management of congestive heart failure. J Am Diet Assoc. 1995 May;95(5):541-4. doi: 10.1016/S0002-8223(95)00148-4. PMID 7722187
- [Background] Pfitzenmeyer P, Guilland JC, d'Athis P, Petit-Marnier C, Gaudet M. Thiamine status of elderly patients with cardiac failure including the effects of supplementation. Int J Vitam Nutr Res. 1994;64(2):113-8. PMID 7960489
- [Background] Falder S, Silla R, Phillips M, Rea S, Gurfinkel R, Baur E, Bartley A, Wood FM, Fear MW. Thiamine supplementation increases serum thiamine and reduces pyruvate and lactate levels in burn patients. Burns. 2010 Mar;36(2):261-9. doi: 10.1016/j.burns.2009.04.012. Epub 2009 Jun 6. PMID 19501976
- [Background] Hung SC, Hung SH, Tarng DC, Yang WC, Chen TW, Huang TP. Thiamine deficiency and unexplained encephalopathy in hemodialysis and peritoneal dialysis patients. Am J Kidney Dis. 2001 Nov;38(5):941-7. doi: 10.1053/ajkd.2001.28578. PMID 11684545
- [Background] Bukhari FJ, Moradi H, Gollapudi P, Ju Kim H, Vaziri ND, Said HM. Effect of chronic kidney disease on the expression of thiamin and folic acid transporters. Nephrol Dial Transplant. 2011 Jul;26(7):2137-44. doi: 10.1093/ndt/gfq675. Epub 2010 Dec 13. PMID 21149507
- [Background] Huertas-Gonzalez N, Hernando-Requejo V, Luciano-Garcia Z, Cervera-Rodilla JL. Wernicke's Encephalopathy, Wet Beriberi, and Polyneuropathy in a Patient with Folate and Thiamine Deficiency Related to Gastric Phytobezoar. Case Rep Neurol Med. 2015;2015:624807. doi: 10.1155/2015/624807. Epub 2015 Nov 30. PMID 26697247
- [Background] Suter PM, Haller J, Hany A, Vetter W. Diuretic use: a risk for subclinical thiamine deficiency in elderly patients. J Nutr Health Aging. 2000;4(2):69-71. PMID 10842416
- [Background] Katta N, Balla S, Alpert MA. Does Long-Term Furosemide Therapy Cause Thiamine Deficiency in Patients with Heart Failure? A Focused Review. Am J Med. 2016 Jul;129(7):753.e7-753.e11. doi: 10.1016/j.amjmed.2016.01.037. Epub 2016 Feb 18. PMID 26899752
- [Background] Crook MA, Sriram K. Thiamine deficiency: the importance of recognition and prompt management. Nutrition. 2014 Jul-Aug;30(7-8):953-4. doi: 10.1016/j.nut.2014.03.003. Epub 2014 Mar 13. No abstract available. PMID 24725734
- [Background] Scheen AJ. Type 2 Diabetes and Thiazide Diuretics. Curr Diab Rep. 2018 Feb 5;18(2):6. doi: 10.1007/s11892-018-0976-6. PMID 29399724
- [Background] Rosenblit PD. Common medications used by patients with type 2 diabetes mellitus: what are their effects on the lipid profile? Cardiovasc Diabetol. 2016 Jul 14;15:95. doi: 10.1186/s12933-016-0412-7. PMID 27417914
- [Background] Jitraknatee J, Ruengorn C, Nochaiwong S. Prevalence and Risk Factors of Chronic Kidney Disease among Type 2 Diabetes Patients: A Cross-Sectional Study in Primary Care Practice. Sci Rep. 2020 Apr 10;10(1):6205. doi: 10.1038/s41598-020-63443-4. PMID 32277150
- [Background] Bailey RA, Wang Y, Zhu V, Rupnow MF. Chronic kidney disease in US adults with type 2 diabetes: an updated national estimate of prevalence based on Kidney Disease: Improving Global Outcomes (KDIGO) staging. BMC Res Notes. 2014 Jul 2;7:415. doi: 10.1186/1756-0500-7-415. PMID 24990184
- [Background] Nazzal Z, Hamdan Z, Masri D, Abu-Kaf O, Hamad M. Prevalence and risk factors of chronic kidney disease among Palestinian type 2 diabetic patients: a cross-sectional study. BMC Nephrol. 2020 Nov 16;21(1):484. doi: 10.1186/s12882-020-02138-4. PMID 33198669
- [Background] Palomares JA, Tummala S, Wang DJ, Park B, Woo MA, Kang DW, St Lawrence KS, Harper RM, Kumar R. Water Exchange across the Blood-Brain Barrier in Obstructive Sleep Apnea: An MRI Diffusion-Weighted Pseudo-Continuous Arterial Spin Labeling Study. J Neuroimaging. 2015 Nov-Dec;25(6):900-5. doi: 10.1111/jon.12288. Epub 2015 Aug 29. PMID 26333175
- [Background] Wu WC, Fernandez-Seara M, Detre JA, Wehrli FW, Wang J. A theoretical and experimental investigation of the tagging efficiency of pseudocontinuous arterial spin labeling. Magn Reson Med. 2007 Nov;58(5):1020-7. doi: 10.1002/mrm.21403. PMID 17969096
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Sanchez-Rangel E, Gunawan F, Jiang L, Savoye M, Dai F, Coppoli A, Rothman DL, Mason GF, Hwang JJ. Reversibility of brain glucose kinetics in type 2 diabetes mellitus. Diabetologia. 2022 May;65(5):895-905. doi: 10.1007/s00125-022-05664-y. Epub 2022 Mar 5. PMID 35247067
- [Background] Gregg JA, Callaghan GM, Hayes SC, Glenn-Lawson JL. Improving diabetes self-management through acceptance, mindfulness, and values: a randomized controlled trial. J Consult Clin Psychol. 2007 Apr;75(2):336-43. doi: 10.1037/0022-006X.75.2.336. PMID 17469891
- [Background] Huang CY, Lai HL, Chen CI, Lu YC, Li SC, Wang LW, Su Y. Effects of motivational enhancement therapy plus cognitive behaviour therapy on depressive symptoms and health-related quality of life in adults with type II diabetes mellitus: a randomised controlled trial. Qual Life Res. 2016 May;25(5):1275-83. doi: 10.1007/s11136-015-1165-6. Epub 2015 Oct 26. PMID 26497665
- [Background] Petrak F, Herpertz S, Albus C, Hermanns N, Hiemke C, Hiller W, Kronfeld K, Kruse J, Kulzer B, Ruckes C, Zahn D, Muller MJ. Cognitive Behavioral Therapy Versus Sertraline in Patients With Depression and Poorly Controlled Diabetes: The Diabetes and Depression (DAD) Study: A Randomized Controlled Multicenter Trial. Diabetes Care. 2015 May;38(5):767-75. doi: 10.2337/dc14-1599. Epub 2015 Feb 17. PMID 25690005
- [Background] Castronovo V, Scifo P, Castellano A, Aloia MS, Iadanza A, Marelli S, Cappa SF, Strambi LF, Falini A. White matter integrity in obstructive sleep apnea before and after treatment. Sleep. 2014 Sep 1;37(9):1465-75. doi: 10.5665/sleep.3994. PMID 25142557
- [Background] Kumar R, Delshad S, Macey PM, Woo MA, Harper RM. Development of T2-relaxation values in regional brain sites during adolescence. Magn Reson Imaging. 2011 Feb;29(2):185-93. doi: 10.1016/j.mri.2010.08.006. Epub 2010 Oct 8. PMID 20933351
- [Background] Kumar R, Delshad S, Woo MA, Macey PM, Harper RM. Age-related regional brain T2-relaxation changes in healthy adults. J Magn Reson Imaging. 2012 Feb;35(2):300-8. doi: 10.1002/jmri.22831. Epub 2011 Oct 10. PMID 21987489
- [Background] Kumar R, Chavez AS, Macey PM, Woo MA, Harper RM. Brain axial and radial diffusivity changes with age and gender in healthy adults. Brain Res. 2013 May 28;1512:22-36. doi: 10.1016/j.brainres.2013.03.028. Epub 2013 Mar 30. PMID 23548596
- [Background] Kumar R, Nguyen HD, Macey PM, Woo MA, Harper RM. Regional brain axial and radial diffusivity changes during development. J Neurosci Res. 2012 Feb;90(2):346-55. doi: 10.1002/jnr.22757. Epub 2011 Sep 21. PMID 21938736
- [Background] Standards of Medical Care in Diabetes-2016: Summary of Revisions. Diabetes Care. 2016 Jan;39 Suppl 1:S4-5. doi: 10.2337/dc16-S003. No abstract available. PMID 26696680
- [Background] American Diabetes Association. Standards of medical care in diabetes-2015 abridged for primary care providers. Clin Diabetes. 2015 Apr;33(2):97-111. doi: 10.2337/diaclin.33.2.97. No abstract available. PMID 25897193
- [Background] Schulz KF, Grimes DA. Unequal group sizes in randomised trials: guarding against guessing. Lancet. 2002 Mar 16;359(9310):966-70. doi: 10.1016/S0140-6736(02)08029-7. PMID 11918933
- [Background] Kumar R, Macey PM, Cross RL, Woo MA, Yan-Go FL, Harper RM. Neural alterations associated with anxiety symptoms in obstructive sleep apnea syndrome. Depress Anxiety. 2009;26(5):480-91. doi: 10.1002/da.20531. PMID 18828142
- [Background] Yadav SK, Kumar R, Macey PM, Woo MA, Yan-Go FL, Harper RM. Insular cortex metabolite changes in obstructive sleep apnea. Sleep. 2014 May 1;37(5):951-8. doi: 10.5665/sleep.3668. PMID 24790274
- [Background] Macey PM, Kumar R, Yan-Go FL, Woo MA, Harper RM. Sex differences in white matter alterations accompanying obstructive sleep apnea. Sleep. 2012 Dec 1;35(12):1603-13. doi: 10.5665/sleep.2228. PMID 23204603
- [Background] Macey PM, Kumar R, Woo MA, Yan-Go FL, Harper RM. Heart rate responses to autonomic challenges in obstructive sleep apnea. PLoS One. 2013 Oct 23;8(10):e76631. doi: 10.1371/journal.pone.0076631. eCollection 2013. PMID 24194842
- [Background] Macey PM, Woo MA, Kumar R, Cross RL, Harper RM. Relationship between obstructive sleep apnea severity and sleep, depression and anxiety symptoms in newly-diagnosed patients. PLoS One. 2010 Apr 16;5(4):e10211. doi: 10.1371/journal.pone.0010211. PMID 20419135
- [Background] Kumar R, Farahvar S, Ogren JA, Macey PM, Thompson PM, Woo MA, Yan-Go FL, Harper RM. Brain putamen volume changes in newly-diagnosed patients with obstructive sleep apnea. Neuroimage Clin. 2014 Jan 31;4:383-91. doi: 10.1016/j.nicl.2014.01.009. eCollection 2014. PMID 24567910
- [Background] Pike NA, Poulsen MK, Woo MA. Validity of the Montreal Cognitive Assessment Screener in Adolescents and Young Adults With and Without Congenital Heart Disease. Nurs Res. 2017 May/Jun;66(3):222-230. doi: 10.1097/NNR.0000000000000192. PMID 28448372
- [Background] Pike NA, Roy B, Gupta R, Singh S, Woo MA, Halnon NJ, Lewis AB, Kumar R. Brain abnormalities in cognition, anxiety, and depression regulatory regions in adolescents with single ventricle heart disease. J Neurosci Res. 2018 Jun;96(6):1104-1118. doi: 10.1002/jnr.24215. Epub 2018 Jan 6. PMID 29315714
- [Background] Singh S, Kumar R, Roy B, Woo MA, Lewis A, Halnon N, Pike N. Regional brain gray matter changes in adolescents with single ventricle heart disease. Neurosci Lett. 2018 Feb 5;665:156-162. doi: 10.1016/j.neulet.2017.12.011. Epub 2017 Dec 6. PMID 29222023
- [Background] Shao X, Ma SJ, Casey M, D'Orazio L, Ringman JM, Wang DJJ. Mapping water exchange across the blood-brain barrier using 3D diffusion-prepared arterial spin labeled perfusion MRI. Magn Reson Med. 2019 May;81(5):3065-3079. doi: 10.1002/mrm.27632. Epub 2018 Dec 18. PMID 30561821
- [Background] Donnino MW, Andersen LW, Chase M, Berg KM, Tidswell M, Giberson T, Wolfe R, Moskowitz A, Smithline H, Ngo L, Cocchi MN; Center for Resuscitation Science Research Group. Randomized, Double-Blind, Placebo-Controlled Trial of Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. Crit Care Med. 2016 Feb;44(2):360-7. doi: 10.1097/CCM.0000000000001572. PMID 26771781
- [Background] Nishimoto A, Usery J, Winton JC, Twilla J. High-dose Parenteral Thiamine in Treatment of Wernicke's Encephalopathy: Case Series and Review of the Literature. In Vivo. 2017 Jan 2;31(1):121-124. doi: 10.21873/invivo.11034. PMID 28064230
- [Background] Madl C, Kranz A, Liebisch B, Traindl O, Lenz K, Druml W. Lactic acidosis in thiamine deficiency. Clin Nutr. 1993 Apr;12(2):108-11. doi: 10.1016/0261-5614(93)90060-h. PMID 16843296
- [Background] Costantini A, Pala MI. Thiamine and fatigue in inflammatory bowel diseases: an open-label pilot study. J Altern Complement Med. 2013 Aug;19(8):704-8. doi: 10.1089/acm.2011.0840. Epub 2013 Feb 4. PMID 23379830
- [Background] Latt N, Dore G. Thiamine in the treatment of Wernicke encephalopathy in patients with alcohol use disorders. Intern Med J. 2014 Sep;44(9):911-5. doi: 10.1111/imj.12522. PMID 25201422
- [Background] Cook CC. Prevention and treatment of Wernicke-Korsakoff syndrome. Alcohol Alcohol Suppl. 2000 May-Jun;35(1):19-20. doi: 10.1093/alcalc/35.supplement_1.19. PMID 11304070
- [Background] Thomson AD, Cook CC. Parenteral thiamine and Wernicke's encephalopathy: the balance of risks and perception of concern. Alcohol Alcohol. 1997 May-Jun;32(3):207-9. doi: 10.1093/oxfordjournals.alcalc.a008259. PMID 9199720
- [Background] Thomson AD, Cook CC, Touquet R, Henry JA; Royal College of Physicians, London. The Royal College of Physicians report on alcohol: guidelines for managing Wernicke's encephalopathy in the accident and Emergency Department. Alcohol Alcohol. 2002 Nov-Dec;37(6):513-21. doi: 10.1093/alcalc/37.6.513. PMID 12414541
- [Background] Wrenn KD, Murphy F, Slovis CM. A toxicity study of parenteral thiamine hydrochloride. Ann Emerg Med. 1989 Aug;18(8):867-70. doi: 10.1016/s0196-0644(89)80215-x. PMID 2757284
- [Background] Kumar R, Ahdout R, Macey PM, Woo MA, Avedissian C, Thompson PM, Harper RM. Reduced caudate nuclei volumes in patients with congenital central hypoventilation syndrome. Neuroscience. 2009 Nov 10;163(4):1373-9. doi: 10.1016/j.neuroscience.2009.07.038. Epub 2009 Jul 24. PMID 19632307
- [Background] Kumar R, Nguyen HD, Ogren JA, Macey PM, Thompson PM, Fonarow GC, Hamilton MA, Harper RM, Woo MA. Global and regional putamen volume loss in patients with heart failure. Eur J Heart Fail. 2011 Jun;13(6):651-5. doi: 10.1093/eurjhf/hfr012. Epub 2011 Mar 9. PMID 21393297
- [Background] Tsai JC, Chen CW, Chu H, Yang HL, Chung MH, Liao YM, Chou KR. Comparing the Sensitivity, Specificity, and Predictive Values of the Montreal Cognitive Assessment and Mini-Mental State Examination When Screening People for Mild Cognitive Impairment and Dementia in Chinese Population. Arch Psychiatr Nurs. 2016 Aug;30(4):486-91. doi: 10.1016/j.apnu.2016.01.015. Epub 2016 Jan 21. PMID 27455923
- [Background] Steer RA, Brown GK, Beck AT, Sanderson WC. Mean Beck Depression Inventory-II scores by severity of major depressive episode. Psychol Rep. 2001 Jun;88(3 Pt 2):1075-6. doi: 10.2466/pr0.2001.88.3c.1075. PMID 11597055
- [Background] Carney CE, Moss TG, Harris AL, Edinger JD, Krystal AD. Should we be anxious when assessing anxiety using the Beck Anxiety Inventory in clinical insomnia patients? J Psychiatr Res. 2011 Sep;45(9):1243-9. doi: 10.1016/j.jpsychires.2011.03.011. Epub 2011 Apr 12. PMID 21482427
- [Background] Beck, A.T. & Steer, R.A. Manual for the Beck Anxiety Inventory. San Antonio, TX: Psychological Corporation: 1993.
- [Background] American Diabetes Association. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S61-S70. doi: 10.2337/dc19-S006. PMID 30559232
- [Background] Ashburner J, Friston KJ. Unified segmentation. Neuroimage. 2005 Jul 1;26(3):839-51. doi: 10.1016/j.neuroimage.2005.02.018. Epub 2005 Apr 1. PMID 15955494
- [Background] Pike, N.A., Woo, M.A., Poulsen, M.K., Halnon, N.J., Lewis, A.B. & Kumar, R. Cognitive impairment in adolescents with congenital heart disease. American Heart Association Annual Meeting, November 15-19, Chicago, IL: 2014.
- [Background] Hollingshead, A.B. Four factor index of social status. New Haven, CT: Yale University Press: 1975.
- [Background] Wiley KD, Gupta M. Vitamin B1 (Thiamine) Deficiency. 2023 Jul 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537204/ PMID 30725889
- [Background] Sullivan EV, Fama R. Wernicke's encephalopathy and Korsakoff's syndrome revisited. Neuropsychol Rev. 2012 Jun;22(2):69-71. doi: 10.1007/s11065-012-9205-2. Epub 2012 May 16. No abstract available. PMID 22588370
- [Background] Thomson, A.D., Guerrini, I. & Marshall, E.J. Wernicke's encephalopathy: role of thiamine. Pract Gastroenterol 33: 21-30, 2009.
- [Background] Crook, M.A. Chapter 6 - Methods for assessment of Thiamine (Vitamin B1). In: Harrington D, editor. Laboratory Assessment of Vitamin Status: Academic Press; 2019. p. 149-64.
- [Background] Owen, A.M., Lee, A.C.H. & Williams, E.J. Dissociating aspects of verbal working memory within the human frontal lobe: Further evidence for a "process-specific" model of lateral frontal organization. Psychobiology 28: 146-55, 2000.
- [Background] Amaral, D.G. & Witter, M.P. Hippocampal formation In: Pacinos G, editor. The rat nervous system. 2nd ed. San Diego, CA Academic Press; 1995. p. 443-93.
- [Background] American Diabetes Association Fast Facts, 2015.
- [Background] Sheslow, D., Adams, W. Wide range assessment of memory and learning administration and technical manual (2nd ed.). Wilmington, DE: Wide Range Inc.; 2003.
- [Background] Beck, A., Steer, R. & Brown, G. Manual for the Beck Depression Inventory-II. San Antonio, Texas: The Psychological Corporation; 1996.
- [Background] Yue, L., Wang, T., Li, G., Li, X., Wang, J., Zhu, M., Li, W. & Xiao, S. Alteration of hippocampus and amygdala in subjective cognitive decline and mild cognitive impairment in community-dwelling chinese. Alzheimer's & Dementia: The Journal of the Alzheimer's Association 13: P405, 2017.
- [Background] Kodl CT, Seaquist ER. Cognitive dysfunction and diabetes mellitus. Endocr Rev. 2008 Jun;29(4):494-511. doi: 10.1210/er.2007-0034. Epub 2008 Apr 24. PMID 18436709
- [Background] Centers for Disease Control and Prevention.National Diabetes Statistics Report: Estimates of diabetes and Its Burden in the United States, 2014. Atlanta, GA: U.S. Department of Health and Human Services; 2014.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT06322212/Prot_ICF_000.pdf